CLINICAL TRIAL: NCT05089838
Title: A Study of CMV-TCR-T Cells in the Treatment of Refractory CMV Viremia After HSCT
Brief Title: CMV-TCR-T Cells for Refractory CMV Infection After HSCT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiao-Jun Huang (Other)
Responsible Party: Sponsor-Investigator, Xiao-Jun Huang, Director, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020PHD014-001
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation; CMV Infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMV-TCR-T cells (Experimental): Patients who enrolled will receive one dose of CMV-TCR-T cells. The dosage ranges from 0.3×10^6 to 1×10^7 TCR+T/Kg.
  Interventions: Biological: CMV-TCR-T cells

INTERVENTIONS:
Biological: CMV-TCR-T cells — Patients who developed refractory CMV infection after allo-HSCT will be enrolled, and donor derived CMV-TCR-T(HLA-A*1101\0201\2402) cells will be intravenously infused with a escalated dose of 0.3-1×10E7CMV-TCR-T cells. The CMV DNA copies and CMV-TCR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14,day 28).

SUMMARY:
This is a single centre, single arm, open-label, phase I study to evaluate the safety and effectiveness of CMV-TCR-T cell immunotherapy in treating refractory CMV infection after HSCT.

DETAILED DESCRIPTION:
CMV infection is a major and potentially life-threatening complication after allogenic hematopoietic stem cell transplantation (allo-SCT). Pharmacotherapy with ganciclovir and foscarnet remains the mainstay of treatment and has significantly improve clinical results, however, it is unsatisfactory owing to toxicity, limited efficacy and risk of developing resistance.

In recent years, adoptive T cell therapy has been proposed as an alternative option for CMV infection after allo-SCT. However, patients with transplants from CMV-negative donors are at highest risk, and an adoptive therapy is missing because CMV-specific T cells are not available.

CMV TCR-transduced donor-derived T Cells (CMV-TCR-T cells) is an attractive strategy to specifically redirect T-cell immunity toward CMV. In this prospective clinical phase I trial, we propose to evaluate the safety and efficacy of stem cell donor-derived CMV-TCR-T cells for patients with refractory CMV infection after allo-SCT. Donor derived CMV-TCR-T(HLA-A*1101\0201\2402) cells will be intravenously infused with a escalated dose of 0.3-1×10E7CMV-TCR-T cells. The CMV DNA copies and CMV-TCR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14, day 28).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute leukemia (AL) or myelodysplastic syndrome (MDS) who receive haploid allogeneic hematopoietic stem cell transplantation, pre-transplantation assessment ≤CR2;
2. Age 18-60, including boundary value, gender unlimited;
3. Refractory CMV infection occurred in the early stage of transplantation : After 2 weeks of standard antiviral treatment, the CMV DNA copy number continued to be ≥1000 copies/mL, and the CMV DNA copy number at the beginning of the treatment decreased by <log10 ；
4. The transplant donor's HLA-A matching is one of 2402, 0201 or 1101, and the physical examination is qualified;
5. ECOG ≤ 3, estimated life expectancy> 3 months;
6. Patients who voluntarily sign informed consent and are willing to comply with treatment plans, visit arrangements, laboratory tests and other research procedures.

Exclusion Criteria:

1. Patients with active aGVHD III-IV and / or mild and severe cGVHD;
2. Have received cell therapy such as DLI, CTL, CAR-T, NK or participated in any other clinical research on drugs and medical devices;
3. Patients who have developed CMV disease;
4. patients with organ failure:

   * Heart: NYHA heart function grade IV;
   * Liver: Grade C that achieves Child-Turcotte liver function grading;
   * Kidney: kidney failure and uremia;
   * Lung: symptoms of respiratory failure;
   * Brain: a person with a disability;
5. Pregnant or lactating women;
6. The researchers found that it was unsuitable for the recipients to be enrolled.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-01-06 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 3 months
  Percentage of participants with adverse events

SECONDARY OUTCOMES:
Changes of CMV-DNA copies | 3 months
  Changes of CMV-DNA copies
CMV-specific immunity reconstitution | 3 months
  In vivo persistence of the infused CMV-TCR-T cells and reconstitution of CMV-specific immunity

CONTACTS AND LOCATIONS:
Overall Officials: Lanping Xu, PhD,MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology,People's hospital Peking University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No